CLINICAL TRIAL: NCT04675996
Title: Phase I/Ib, Open-label, Multiple Ascending Dose, First-in-Human Study, to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of INT-1B3 in Patients With Advanced Solid Tumors
Brief Title: First-in-Human Study of INT-1B3 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: insufficient funding
Sponsor: InteRNA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT1B3-CLIN-101
Record Dates: First submitted 2020-12-08; First posted 2020-12-19 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor
Keywords: MicroRNA; Solid Tumor; Lipid-nanoparticle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase 1/1b (Experimental): Phase 1: dose escalation phase with a 'hybrid' 3+3 design in all-comers cancer patients. Approximately 30 patients will be included.
  Phase 1b: dose expansion phase in selected tumor types at the recommended phase 2 dose. Approximately 50 patients will be included.
  Interventions: Drug: INT-1B3

INTERVENTIONS:
Drug: INT-1B3 — 60-min i.v. infusions twice per week in 21-day cycles

SUMMARY:
This is a 2 part, multi-center, open-label, First-in-Human clinical study to evaluate the safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of INT-1B3 in the treatment of patients with advanced solid tumors.

DETAILED DESCRIPTION:
The investigational medicinal product INT-1B3 is a lipid nanoparticle formulated microRNA (miR-193a-3p) mimic destined for therapeutic intervention in oncology. Preclinical work showed that INT-1B3 has a multi-target mechanism of action with an anti-proliferative, anti-metastatic, anti-migration, cell cycle disruption, induction of apoptosis effect and modulation on the tumor microenvironment leading to significant induction of T cell-mediated immune response.

The first part of the study (Phase I) is a dose-escalation phase to determine the maximal tolerated dose and the recommended Phase 2 dose, as well as the safety profile of INT-1B3 in patients with advanced malignancies.The subsequent expansion phase of the study (Phase Ib) will further explore safety, pharmacokinetics, pharmacodynamic responses, and antitumor activity of INT-1B3 in patients with selected cancer types treated at the recommended phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

1. Patient provided a signed written informed consent before any screening procedure
2. Patient is male or female, ≥18 years of age (adult patients)
3. Patient with histologically or cytologically confirmed advanced and/or metastatic solid tumor, with progressive disease at baseline, for whom no standard treatment is available or who have declined standard therapy
4. Patient with evaluable disease per RECIST v1.1, iRECIST
5. Patient with a predicted life expectancy of > 12 weeks
6. Patient with Eastern Cooperative Oncology Group performance status of grade 0 - 1
7. Patient with hemoglobin ≥ 9.0 g/dL, platelet count ≥ 75×109/L, and absolute neutrophil count ≥ 1.0×109/L
8. Patient with adequate renal function
9. Patient with adequate liver function
10. Patient with adequate coagulation tests
11. Female patient of childbearing potential and males should use effective contraception
12. Patient is able and willing to comply with the protocol and the restrictions and assessments therein

Exclusion Criteria:

1. Patients on any other anti-cancer therapy, unless at least 4 weeks (or 5 half-lives, whichever is shorter), have elapsed since the last dose before the first administration of INT-1B3. At least 2 weeks should have elapsed since receiving non-palliative radiotherapy.
2. Patient with known central nervous system (CNS) metastases, unless previously treated and well-controlled for at least 1 month (defined as clinically stable, no edema, no steroids and stable in 2 scans at least 4 weeks apart)
3. Patient with concomitant second malignancies unless curatively treated at least 2 years before study entry with no additional therapy required or anticipated to be required during the study period
4. Patient with major surgery within 5 weeks before initiating treatment or with minor surgical procedure within 7 days before initiating treatment
5. Patient with active autoimmune disease or persistent immune-mediated toxicity caused by immune checkpoint inhibitor therapy of Grade ≥ 2, except for residual endocrinopathy adequately substituted, vitiligo, Type 1 diabetes mellitus or psoriasis not requiring systemic therapy (>10mg prednisone equivalent)
6. Patient with toxicity (except for alopecia) related to prior anti-cancer therapy and/or surgery, unless the toxicity is either resolved, returned to baseline or grade 1
7. Patient with any active neuropathy > Grade 2 (National Cancer Institute Common Terminology Criteria for Adverse Events v5.0)
8. Patient with any condition requiring concurrent use of systemic immunosuppressants or corticosteroids at a daily dose > 10 mg prednisone equivalent or other immunosuppressive medications within 14 days of study medication administration
9. Patient with evidence of active infection that requires systemic antibacterial, antiviral, or antifungal therapy ≤ 7 days before the first dose of study medication
10. Patient with uncontrolled or significant cardiovascular disease
11. Patient with known active or chronic hepatitis B or C (unless treated with no detectable virus)
12. Patient with known history of exposure to human immunodeficiency virus (HIV)
13. Patient with any known or underlying medical, psychiatric condition, and/or social situations that, in the opinion of the investigator, would limit compliance with study requirements
14. Patient with history of allergy to the study medication or any of its excipients
15. Patient that received packed red blood cells or platelet transfusion within 2 weeks of the first dose of study medication
16. Female patient: pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-related adverse events and serious adverse events | Up to 24 months
  Incidence and severity of adverse events, serious adverse events, according to NCI-CTCAE criteria v 5.0, incidence of dose limiting toxicities (DLTs), adverse events leading to discontinuation and deaths
Recommended Phase 2 Dose of INT-1B3 | Up to 24 months
  Based on dose-limiting toxicities, the maximal tolerated dose and all other available safety, pharmacokinetic/pharmacodynamic data as assessed by the cohort review committee

SECONDARY OUTCOMES:
Area under the curve | Up to 24 months
  Area under the plasma concentration time curve of INT-1B3
Maximum plasma concentration | Up to 24 months
  Highest observed plasma concentration of INT-1B3
Time of maximum plasma concentration | Up to 24 months
  Time to reach highest observed plasma concentration of INT-1B3
Half-life | Up to 24 months
  Plasma concentration half-life of INT-1B3
Objective response rate of INT-1B3 | Up to 24 months
  Objective response rate according to standard criteria by RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Roel Schaapveld, PhD, Study Director — InteRNA
Locations (4):
- Belgium (2):
  - Institut Jules Bordet, Brussels, Wallonia
  - GZA (Gasthuiszusters Antwerpen), Antwerp
- Netherlands (2):
  - The Netherlands Cancer Institute, Amsterdam
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: No